CLINICAL TRIAL: NCT07309458
Title: Effectiveness of a Nursing Intervention on Pre-surgical Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Elena Violeta Iborra Palau, Principal Investigator, University of Valencia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024.044
Record Dates: First submitted 2025-12-15; First posted 2025-12-30 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Pre Surgical Anxiety
Keywords: pre surgical anxiety; Nursing intervention
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: Experimental study with a control group of nursing intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Control Group without nursgin intervention
- Intervention (Experimental): Intervention Group with nursing intervention
  Interventions: Behavioral: Nursing Intervention

INTERVENTIONS:
Behavioral: Nursing Intervention — Specific Nursing Intervención to reduce pre surgical anxiety based on Nursing Intervention Taxonomy (NIC)
  Arms: Intervention

SUMMARY:
Preoperative anxiety is a very common experience among surgical patients. Many people scheduled for Day Surgery (Ambulatory Major Surgery, AMS) experience worry, tension, or fear while waiting to enter the operating room. This anxiety is not incidental; numerous studies have shown that it can influence pain perception, postoperative recovery, and overall satisfaction with the surgical procedure. Despite its relevance, routine clinical practice does not always include structured interventions to help patients manage these feelings in the moments immediately before surgery. Due to their close and continuous role throughout the surgical process, nursing professionals are key in providing this type of support.

This clinical study is being conducted at Hospital de la Malvarrosa (Valencia) and focuses on adult patients scheduled for AMS across different surgical specialties, including Otorhinolaryngology, Maxillofacial Surgery, General Surgery, and Urological Surgery. Its aim is to provide a clear, evidence-based answer to the following question: can an individualized nursing intervention applied in the immediate preoperative period reduce anxiety levels and improve the patient's overall surgical experience? The study hypothesis proposes that a brief, personalized intervention delivered by nursing staff-based on empathic communication, tailored information, and simple coping techniques-can help patients manage preoperative anxiety and positively influence their perception of the surgical process.

To test this hypothesis, the study compares two groups of patients undergoing AMS. The control group receives standard preoperative care, which includes clinical preparation and the basic information routinely provided before surgery. The intervention group, in contrast, receives an additional individualized nursing intervention lasting approximately 15-20 minutes in the preoperative area, carried out alongside routine preparation procedures such as intravenous cannulation, medication administration, or surgical checklist verification. During this process, the nurse creates a trusting environment, encourages patients to express their fears, validates their emotions, provides clear and understandable explanations of the different stages of the procedure, and teaches simple breathing and emotional regulation techniques.

Anxiety levels are assessed using a validated clinical scale that measures both physical and emotional symptoms related to anxiety. Assessment takes place in the immediate preoperative period, allowing for an objective comparison between the control and intervention groups. In addition, the study collects data on personal, social, and surgical variables that may influence anxiety, with the aim of better understanding which patient profiles are more vulnerable and which benefit most from the intervention.

Although the primary approach of the study is quantitative, a qualitative perspective is also incorporated to explore the subjective experiences of both patients and nursing staff.

Overall, this study aims to demonstrate that a humanized, structured, and evidence-based nursing intervention can significantly reduce preoperative anxiety in AMS and improve the surgical experience. Furthermore, it seeks to contribute knowledge that supports the development of more comprehensive care protocols in which patients' emotional well-being is considered an essential component of surgical preparation.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old.
* Voluntary participation and informed consent to participate in the study.
* Individuals scheduled for major outpatient surgical procedures in operating rooms 5 and 6 of La Malvarrosa Hospital

Exclusion Criteria:

* Patients with comprehension difficulties (hearing loss, language barrier, or insufficient cognitive level).
* Patients with temporarily impaired cognitive ability (premedicated with benzodiazepines)
* Clinical situations that prevented participation in data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Change in Anxiety Severity assessed by the Hamilton Anxiety Rating Scale (HAM-A) | Baseline (upon a arrival at holding area) and inmediatly post nursing intervention (approximately 20 minutes after baseline)
  The HAM-A consists of 14 items that measure both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Each item is scored on a scale of 0 (not present) to 4 (very severe). The total score ranges from 0 to 56, obtained by summing the scores of all 14 items. Higher scores indicate higher levels of anxiety (worse outcome). Scores are interpreted as follows: 0-17 (mild anxiety), 18-24 (moderate anxiety), 25-30 (severe anxiety), and >30 (very severe anxiety).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Malvarrosa, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
The anonymized database from the study will be shared via the Zenodo platform. Initially, the data will remain hidden and will only be shared once the study has been published.